CLINICAL TRIAL: NCT05914038
Title: Efficacy of Individualized Repetitive Transcranial Magnetic Stimulation Based on Cortical Laterality for Motor Recovery in Stroke Patients
Brief Title: Individualized rTMS for Motor Recovery in Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202301225DIND
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Stroke; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- individualized rTMS (Experimental): Patients will receive individualized repetitive transcranial magnetic stimulation according to lateralization index measured by functional near-infrared spectroscopy
  Interventions: Device: Repetitive transcranial magnetic stimulation
- Traditional rTMS (Active Comparator): Control group is given traditional rTMS
  Interventions: Device: Repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive neuromodulation technology. High and low frequencies of rTMS could modulate the excitability of the cerebral cortex.

SUMMARY:
This study aimed to aim to investigate the efficacy of individualized rTMS according to lateralization index on motor recovery and cortical excitability in subacute stroke patients.

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive neuromodulation technology.

High and low frequencies of rTMS could modulate the excitability of the cerebral cortex. Theta burst stimulation (TBS) has achieved a similar effect to traditional rTMS mode.

However, the current rTMS studies for stroke patients utilized the same therapeutic protocol and there is no individualized rTMS protocol based on the value of lateralization index.

This study aimed to aim to investigate the efficacy of individualized rTMS according to lateralization index on motor recovery and cortical excitability in subacute stroke patients.

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral ischemic or hemorrhagic stroke
2. Stroke within 3 months
3. Medical Research Council Scale for Muscle Strength in upper limb ≤ 3
4. No previous stroke, seizure, dementia, Parkinson's disease or other degenerative neurological diseases.
5. Patient could sit over 15 minutes
6. Age over 20

Exclusion Criteria:

1. Previous stroke, traumatic brain injury, brain tumor
2. With central nervous system disease (spinal cord injury, Parkinson's disease)
3. Any contraindication to rTMS (seizure, alcoholism, metal implant, pacemaker)
4. Patients unable to cooperate the treatment
5. Pregnancy
6. Depression

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-13 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2027-05-20 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment | 12 weeks post intervention
  Fugl-Meyer Assessment motor function set, score: 0-66, higher scores indicate a better outcome.

SECONDARY OUTCOMES:
Medical Research Council (MRC) Scale for Muscle Strength | 1 week, 4 weeks, 12 weeks post intervention
  Medical Research Council (MRC) Scale for Muscle Strength, assessing muscle strength from Grade 5 (normal) to Grade 0 (no visible contraction).
National Institutes of Health Stroke Scale | 1 week, 4 weeks, 12 weeks post intervention
  National Institutes of Health Stroke Scale, The maximum possible score is 42, with the minimum score being a 0. Higher scores indicate a worse outcome.
Barthel Index | 1 week, 4 weeks, 12 weeks post intervention
  Barthel Index, score 100-0. Higher scores indicate a better outcome.
Modified Rankin Scale | 1 week, 4 weeks, 12 weeks post intervention
  Modified Rankin Scale, score from 0 to 6. Higher scores indicate a worse outcome.
MEP | 1 week, 4 weeks, 12 weeks post intervention
  motor evoked potential
Fugl-Meyer Assessment | 1 week, 4 weeks post intervention
  Fugl-Meyer Assessment motor function set, score: 0-66, higher scores indicate a better outcome.
functional NIRS | 1 week, 4 weeks, 12 weeks post intervention
  Functional Near Infrared Spectroscopy to detect the cortical excitability

CONTACTS AND LOCATIONS:
Overall Officials: Meng Ting Lin, M.D., Principal Investigator — The Department of Physical Medicine and Rehabilitation, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei County, Taipei, Taiwan